CLINICAL TRIAL: NCT07127250
Title: Interest of Walking Sticks to Increase Walking Activity of People With Sagittal Imbalance of Spine: a Comparative Exploratory Study (Before-after) Using Mixed Methodology.
Brief Title: Interest of Walking Sticks to Increase Walking Activity of People With Sagittal Imbalance of Spine
Acronym: WALKSPINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP250475; IDRCB (Registry Identifier: 2025-A00608-41)
Record Dates: First submitted 2025-07-16; First posted 2025-08-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Static Spinal Disorder
Keywords: Walking sticks; Walking distance; Static spinal disorder; Spinal static disorder; Anterior imbalance of spine; Pedometer
MeSH Terms: interventions — Canes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking sticks (Experimental)
  Interventions: Other: Walking sticks

INTERVENTIONS:
Other: Walking sticks — Walking with walking sticks and pedometer Daily walking activity recorded in a logbook

SUMMARY:
The purpose of this pilot study is to assess the impact of using walking sticks on walking perimeter in people with anterior spinal imbalance.

DETAILED DESCRIPTION:
Aging is associated with a number of highly prevalent spinal pathologies, characterized by static disorders affecting spinal balance in the sagittal plane especially. These postural disorders are a source of pain, activity limitation and reduced quality of life. Treatment of spinal static disorders is essentially symptomatic based on medical care and rehabilitation and includes the use of spinal orthosis. Adherence to spinal orthosis is poor.

Walking requires dynamic stabilization capacities, which are affected by static disorders of the spine. In the case of walking difficulties associated with sagittal imbalance of spine, the walking aid most frequently assessed in the literature is the rollator. Using a rollator promotes anterior flexion of the spine and prevents physiological dissociation of the scapular and pelvic girdles.

Walking sticks help maintain sagittal alignment of the spine, improving the subject's dynamic stability while respecting the physiological gait pattern (dissociation of the scapular and pelvic belts).

To date, no study has assessed the impact of using walking sticks to increase walking activity in a population of people with sagittal imbalance of spine.

Deterioration in overall spinal balance and reduced stabilization capabilities are associated with increased risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 50 years
* VAS (Sagittal Vertical Axis, C7-S1, EoS (clinical follow-up)) > 5cm
* Able to do transfers alone
* Able to walk 10 minutes or 400 meters in a row
* Self-reported Walking difficulties
* Person living at home
* Person willing and consenting to participate in the study
* Health insurance

Exclusion Criteria:

* Current use of walking sticks
* Advanced and symptomatic osteoarthritis of the lower limbs
* Static disorder of the fixed spine
* Introduction of a straightening brace in the 3 months preceding the start of the study
* Static disorder explained by infectious, tumoral, congenital or neurodegenerative pathologies
* Uncompensated lower-limb length inequality (> 2cm)
* Lower limb motor deficit
* Upper limb pathology preventing cane use
* Proprioceptive or vestibular pathology
* Inability to write, speak or read French
* Cognitive and/or behavioral disorders
* Participation in other research on spinal balance and/or gait, or that could influence these factors during the study period
* People under tutorship or curatorship
* Free state medical assistance

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Walking perimeter | Day 0 and month 3 (+ 15 days, 13 to 15 weeks)
  6-minute walk test at Day 0 without walking sticks and 3 months later with walking sticks

SECONDARY OUTCOMES:
Number of daily steps | Periods Day 1-Day 7 and Day 8-Month 3
  Daily steps measured by pedometer
Walking perimeter | Day 0 and month 3
  6-minute walk test at Day 0 without walking sticks and 3 months later without walking sticks
Postural stability parameters | Day 0 and month 3
  Postural stability parameters (measured on a stabilometry platform, Abilycare).
Spatio-temporal walking parameters | Day 0 and Month 3
  Variation in spatio-temporal walking parameters (measured on a GaitRite treadmill
Number of falls in the last 3 months | Day 0 and Month 3
Mean spinal pain | Day 0 and Month 3
  Variation in the average intensity of spinal pain (in the last 48 hours) (Numerical Scale, 0: no pain, 10: maximum imaginable pain)
Activity limitation | Day 0 and Month 3
  Variation in activity limitation assessed by the self-completed Oswestry Disability Index (ODI, 0-50, no activity limitation; 50 maximum limitation)
Quality of life | Day 0 and Month 3
  Variation in specific quality of life assessed by the Scoliosis Research Society-22 revised self-assessment questionnaire (SRS-22r, for each of the 5 domains, score from 1: minimum quality of life to 5: maximum quality of life).
Participant's opinions on the use of sticks collected | Month 3
  Using open and closed questions

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra ROREN, Study Director — Assistance Publique - Hôpitaux de Paris; Rémy FLECHON, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de rééducation et de réadaptation de l'appareil locomoteur et des pathologies du rachis.Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No